CLINICAL TRIAL: NCT01695902
Title: A Multiple Center, Randomised, Parallel Group, Single-blind Clinical Trial, to Assess the Therapeutic Equivalence in Terms of Efficacy and Safety of Test Product (Levosert) and Reference Product (Mirena®) in Patients With Menorrhagia - Phase III (Therapeutic Equivalence).
Brief Title: Therapeutic Equivalence Trial of Two Hormonal-IUDs in Patients With Heavy Menstrual Bleeding
Acronym: LVS-20
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Uteron Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-001564-77
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levosert-20 (Experimental): Levosert is a LNG-releasing Intrauterine Delivery System (IUS) containing 52 mg of LNG in a cylindrical-shaped reservoir. The reservoir is mounted on the vertical arm of a T-shaped plastic frame and is covered with a release rate controlling membrane.
  Interventions: Drug: Levosert-20
- Mirena® (Active Comparator): Mirena® IUS, Bayer-Schering, a LNG-releasing Intrauterine Delivery System (IUS) containing 52 mg of LNG.
  Interventions: Drug: Mirena

INTERVENTIONS:
Drug: Levosert-20
  Arms: Levosert-20
Drug: Mirena
  Arms: Mirena®

SUMMARY:
The primary objective of this study was to compare the efficacy of Test Product (Levosert) vs. Reference Product (Mirena® Bayer-Schering) based on the mean variation of menstrual blood loss volume in women with menorrhagia.

The secondary objectives includes physical and gynaecological examinations, vital signs, clinical laboratory tests including hemoglobin and ferritin measurements, body weight and spontaneously reported adverse events were analysed and compared between Levosert and Mirena® treatment arms. Plasma levels of levonorgestrel (LNG) were also evaluated after various periods of time. The residual amounts of LNG in the devices were finally measured after withdrawal at completion of the study. Plasma levels of LNG and residual amounts of LNG were compared between the two treatment groups. Contraceptive effect of Levosert was estimated by Pearl Index.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-planning pregnancy, non-lactating non-menopausal females at least 18 years of age.
* Patients with a clinical diagnosis of functional Menorrhagia during the last 6 months.
* Patients who are eligible and able to participate in the trial and who consent to do so in writing after the purpose and nature of the investigation have been explained to them.

Exclusion Criteria:

* History of endometrial ablation or dilatation and/or curettage within the 3 months prior to screening
* Copper - coiled-intrauterine device or LNG releasing IUS use within 2 months prior to screening
* Abnormal liver function or jaundice
* Renal insufficiency
* Other hormonal treatment (sexual steroids),
* Organic causes of abnormal uterine bleeding (presence of endometrial polyps, submucous myomas of any size, or myometrial myomas > than 3 cm, adenomyosis, atypical hyperplasia, carcinoma)
* Abnormal uterine morphology
* Presence of ovarian cyst > 3 cm
* Lower genital tract infection
* Current or recurrent PID (present or recurrent pelvis infection (including history of postpartum endometritis, infected miscarriage) during the past 3 months
* Uncontrolled hypertension
* Congenital or acquired valvular disease (including corrections with prosthetic valves)
* Known or suspected pregnancy
* Known or suspected hormone-dependent tumor
* BMI > 30
* Abnormal Pap smear test or other evidence of cervical/endometrial mancy
* Unexplained amenorrhea
* Known hypersensitivity to device material and/or Levonorgestrel

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Year 1 in the mean menstrual blood loss volume measured using the modified Wyatt pictogram in the two treatment groups | 1 year

SECONDARY OUTCOMES:
Comparison of the plasma levels of LNG (Levonorgestrel) in the 2 treatment groups | up to three years
Comparison of the residual LNG level in the IUS in the 2 treatment groups | up to three years
Mean reduction in menstrual blood loss volume from baseline to intermediate cycles (equivalent to 28-days period) | 1 year

OTHER OUTCOMES:
Change from baseline to year 1/year 3 in weight in the 2 treatment groups | up to three years
Change from baseline to year 1 / year 3 in hemoglobin in the 2 treatment groups | up to three years
Change from baseline to year 1/year 3 in ferritin in the 2 treatment groups | up to three years
Occurrence in the 2 treatment groups of evaluable untoward drug reactions | up to three years
Contraception level and contraceptive effect in the 2 treatment groups | up to three years